CLINICAL TRIAL: NCT07026552
Title: Proteomic and Histological Analysis of Ligamentum Flavum Hypertrophy and Degeneration in Lumbar Spinal Stenosis: Clinical, Surgical, and Therapeutic Implications
Brief Title: Proteomic and Histological Analysis of Ligamentum Flavum in Lumbar Stenosis
Acronym: APIDeLeG
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, La Rocca Giuseppe, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 7092
Record Dates: First submitted 2025-03-07; First posted 2025-06-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Spinal Stenosis of Lumbar Region; Spine Degeneration
Keywords: Lumbar Spinal Stenosis; Ligamentum Flavum Hypertrophy; Proteomic Analysis; Molecular Biomarkers
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ligamentum Flavum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lumbar Spinal Stenosis Surgery Group: This cohort consists of patients undergoing decompression surgery for lumbar spinal stenosis. Tissue and biological fluid samples will be collected intraoperatively to analyze molecular and histological characteristics associated with ligamentum flavum hypertrophy (LFH).
- Other Degenerative Spinal Disease Surgery Group: This cohort includes patients undergoing surgery for other degenerative spinal conditions of the spine such as lumbar disk herniation. Ligamentum flavum samples from this group will serve as a comparative control to assess differences in molecular, histological, and proteomic profiles between non-LFH and LFH tissues.

SUMMARY:
Background Lumbar spinal stenosis (LSS) is a common condition characterized by spinal canal narrowing, often linked to ligamentum flavum hypertrophy (LFH) and degeneration. Fibrotic processes involving elastin and collagen alterations contribute to LF thickening and spinal instability. Despite progress, the molecular mechanisms underlying LFH remain unclear, necessitating targeted diagnostic and therapeutic strategies.

Objective This study aims to analyze the proteomic and histological changes in LFH associated with LSS, correlating molecular signatures with imaging and surgical findings to identify potential therapeutic targets.

Methods LF samples from LSS patients undergoing surgery will be analyzed using mass spectrometry-based proteomics and histology to identify biomarkers and molecular pathways. Correlations between imaging, intraoperative findings, and molecular profiles will be assessed.

Expected Results The study aims to identify specific biomarkers and molecular pathways involved in LFH, linking them to clinical and imaging findings. Statistical analyses will evaluate associations between molecular alterations and surgical outcomes to define therapeutic targets.

Significance By identifying molecular markers of LFH, this research aims to improve LSS diagnosis and treatment, potentially guiding targeted therapies to slow disease progression and enhance patient outcomes.

Study Design A multidisciplinary team from Fondazione Policlinico Universitario Agostino Gemelli and Università Cattolica del Sacro Cuore will conduct the study, ensuring robust data integration and statistical evaluation.

Conclusion This comprehensive study will provide valuable insights into the molecular and histological modifications associated with LFH in LSS, paving the way for new therapeutic approaches to improve patient outcomes and satisfaction.

DETAILED DESCRIPTION:
1. INTRODUCTION Lumbar spinal stenosis (LSS) is a highly prevalent condition worldwide, characterized by the narrowing of the spinal canal. Epidemiological studies indicate a high incidence of LSS, influenced by demographic shifts and the increasing burden of age-related musculoskeletal disorders. The etiology of LSS is primarily classified as acquired (degenerative) or congenital, affecting approximately 103 million individuals globally. The degenerative form becomes increasingly common with advancing age. Anatomically, degenerative LSS is subdivided into central, lateral, and foraminal stenosis, with the highest prevalence observed at the L4-L5 level. Key etiological factors include thickening and deformation of the ligamentum flavum (LF), often resulting from reduced disc height, facet joint hypertrophy, or a combination of both. Among these factors, ligamentum flavum hypertrophy (LFH) is recognized as the primary cause of lumbar spinal canal stenosis (LSCS).

   The LF is a crucial structure connecting the laminae of adjacent vertebrae, composed of approximately 80% elastic fibers and 20% collagen fibers. It plays a vital role in forming the posterior boundary of the spinal canal, preventing excessive flexion of the vertebral column, and maintaining spinal stability. Several studies indicate that individuals with hypertrophic LF exhibit a reduction and disorganization of elastic fibers, accompanied by an increase in collagen fibers, suggesting that LFH is driven by a fibrotic process. Identifying risk factors for LFH remains challenging and is a subject of ongoing debate in the literature; age and mechanical stress are currently considered the most significant contributors.

   Few studies have focused on elucidating the molecular mechanisms underlying LSS and LFH or on identifying specific diagnostic and prognostic biomarkers. As a result, the pathophysiology and molecular basis of LSS and LFH remain poorly understood, underscoring the need for precise molecular characterization and the development of targeted treatments based on specific molecules.

   Zhao et al. identified a significant increase in thrombospondin-1 (THBS1) expression in LFH using proteomics and single-cell RNA sequencing in clinical samples. Laboratory experiments demonstrated that THBS1 activates the Smad3 signaling pathway via transforming growth factor β1 (TGF-β1), enhancing the expression of fibrotic markers COL1A2 and α-SMA. A bipedal murine model confirmed the crucial role of THBS1 in LFH development. Additionally, sestrin2 (SESN2), a stress-responsive protein, was shown to suppress THBS1 expression, preventing fibrosis in LF cells. These findings suggest that mechanical overload increases THBS1 production, triggering the TGF-β1/Smad3 pathway and leading to tissue hypertrophy. Suppressing THBS1 expression could provide a novel therapeutic approach for LFH.

   In another study, Wang et al. found that wild-type amyloid transthyretin (ATTRwt) was present in LF samples from patients undergoing decompression surgery, with amyloid load positively correlating with LF thickness and lumbar LF burden in a dose-dependent manner.

   Liu et al. reported that hypertrophic LF samples exhibited higher levels of CLU, TGF-β1, α-SMA, ALK5, and phosphorylated SMAD3 proteins compared to non-LFH samples. Mechanical stress and TGF-β1 were found to induce clusterin (CLU) expression in LF cells. Notably, CLU inhibited COL1A2 and α-SMA expression, which were stimulated by mechanical stress and TGF-β1. Mechanistic studies demonstrated that CLU suppressed mechanical stress-induced and TGF-β1-driven SMAD3 activity by inhibiting SMAD3 phosphorylation and nuclear translocation through competitive binding with ALK5. Additionally, PRKD3 stabilized CLU protein, preventing its lysosomal degradation. In vivo experiments showed that CLU attenuated LFH induced by mechanical stress. These results suggest that CLU mitigates LFH by modulating TGF-β1 signaling pathways both in vitro and in vivo, acting as a negative feedback regulator of TGF-β1 and inhibiting fibrotic responses in LF.

   Zheng et al. discovered that TGF-β1 significantly increased CRLF1 mRNA expression via the SMAD3 pathway. CRLF1 was found to enhance LF fibrosis through the ERK signaling pathway at the post-transcriptional level and was essential for the pro-fibrotic effects of TGF-β1. When CRLF1 was silenced, fibrosis induced by inflammatory cytokines and mechanical stress was reduced. Furthermore, experiments demonstrated that bipedal posture could induce LFH and increased CRLF1 expression in mice. Overexpression of CRLF1 led to LFH in vivo, whereas CRLF1 silencing prevented LFH development in bipedal mice.

   These studies highlight the critical role of specific molecules in the development and regulation of LFH. However, the pathogenesis remains incompletely elucidated. Further research is required to clarify these mechanisms and develop potential strategies for the prevention and treatment of LFH and LSS.
2. OBJECTIVES AND CLINICAL TRIAL AIMS (HYPOTHESIS AND EXPECTED OUTCOMES) The objective of this study is to conduct a comprehensive clinical and proteomic investigation of LFH, comparing molecular profiles of different LF samples within a well-defined patient cohort that meets inclusion criteria and has a statistically significant sample size. Proteomics is a valuable tool for studying diseases at the molecular level, helping to elucidate mechanisms involved in inflammatory responses and biomechanical stress.

   Specifically, Clinical Proteomics, as applied in this project, focuses on the biomedical application of proteomics and integrates proteomics, epidemiology, clinical chemistry, and medical disciplines, aligning perfectly with the study's objectives. This approach involves determining the total protein expression profile of a specific cell, tissue, or body fluid at a given time, assessing qualitative and quantitative differences between healthy and diseased subjects.

   This project integrates multiple research units, where clinicians, neurosurgeons, biochemists, and molecular biologists collaborate closely to achieve the desired outcomes, each contributing their expertise to the study.
3. STUDY DESIGN

   3.1 Study Type: Prospective, single-center observational study.

   3.2 Study Duration: The study will commence following approval by the Ethics Committee and will last for 36 months.

   3.3 Study Endpoints

   3.3.1 Primary Endpoint

   Investigate molecular and histological aspects through proteomic and microscopic analysis to identify a potential specific pattern in LSS patients, comparing them with a healthy population.

   3.3.2 Secondary Endpoints

   Correlate blood test results (routine clinical blood sampling) with a specific LFH pattern.

   Assess correlations between preoperative imaging findings and intraoperative and molecular results.

   3.4 Experimental Procedures

   Provide a molecular characterization of the ligamentum flavum in two study populations (non-degenerative disease vs. degenerative disease) through the application of an integrated proteomic approach based on top-down and bottom-up platforms. The data could provide valuable insights into the molecular mechanisms underlying the onset and progression of the disease.

   Identify molecular biomarkers for clinical applications: The analysis of different ligamentum flavum samples could reveal specific proteins associated with spinal stenosis and clarify the mechanisms regulating these pathways. The identification of these biomarkers could significantly improve the treatment of lumbar spinal stenosis by introducing new therapeutic targets to mitigate inflammatory and hypertrophic responses, slow stenosis progression, and ultimately enhance patients' quality of life.
4. STUDY POPULATION (SAMPLE SIZE CALCULATION) Patients undergoing decompression surgery for lumbar spinal stenosis will be compared with patients undergoing surgery for other degenerative spinal diseases.
5. DATA ANALYSIS AND SAMPLE SIZE

   5.1 SAMPLE SIZE Given the nature of the study, a formal sample size determination is not required. Based on the number of patients treated annually, we estimate enrolling 100 patients who meet the inclusion and exclusion criteria within 24 months and describing their proteomic patterns. Ligamentum flavum samples will be obtained from 50 patients undergoing decompression surgery for lumbar spinal stenosis and compared with samples from 50 patients undergoing surgery for other degenerative spinal diseases.

   5.2 HISTOLOGICAL ANALYSIS The samples will be stained and examined to detect changes in the composition of collagen and elastin fibers, cellularity, and the presence of inflammatory markers. Advanced imaging techniques will be employed to quantify tissue alterations.

   5.3 MOLECULAR ANALYSIS RNA and protein extracts from ligamentum flavum samples will be analyzed using techniques such as qPCR, Western blotting, and immunohistochemistry to identify gene and protein expression changes related to fibrosis, inflammation, and extracellular matrix remodeling.

   5.4 PROTEOMIC ANALYSIS Ligament samples will undergo proteomic analysis using mass spectrometry platforms, employing integrated top-down and bottom-up approaches.

   5.5 STATISTICAL ANALYSIS Quantitative variables following a normal distribution will be summarized as mean and standard deviation (SD) or, otherwise, as median and interquartile range (IQR).

   Categorical variables will be reported as absolute and relative frequencies (percentage).

   Normality of variables will be assessed using the Shapiro-Wilk test. Comparisons between categorical variables will be performed using the chi-square test or Fisher's exact test.

   Differences between quantitative variables will be tested using Student's t-test or the Mann-Whitney test.

   Preoperative and postoperative clinical data, functional outcomes, and imaging results will be collected and correlated with histological and molecular data to identify potential biomarkers and predictors of surgical outcomes through linear regression analysis.

   Correlation between various parameters will be further evaluated by calculating the Pearson and/or Spearman correlation coefficient.

   Results will be considered statistically significant at p<0.05. Analyses will be conducted using R statistical software (R, CRAN).
6. DIRECT ACCESS TO DATA/ORIGINAL DOCUMENTS The Principal Investigator or their delegates must allow the Regulatory Authority, the Independent Ethics Committee, or the Sponsor (or their delegates) free access and the ability to conduct relevant audits on all original study documentation, including informed consent forms signed by enrolled subjects, relevant medical records, and/or outpatient registers. Individuals granted access to the documentation must take all reasonable precautions to maintain the confidentiality of subject identities in compliance with applicable legislation.
7. GOOD CLINICAL PRACTICE REGULATIONS This study will be conducted in accordance with the principles of Good Clinical Practice (GCP) (Group, 1996), the Declaration of Helsinki, and national regulations governing the conduct of clinical trials. By signing the protocol, the investigator agrees to adhere to the procedures and instructions contained therein and to conduct the study in compliance with GCP, the Declaration of Helsinki, and national laws regulating clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Radiological (CT and/or MRI) and clinical evidence of lumbar spinal stenosis (LSS).
* Age range: 50-85 years.
* Signed informed consent, medical records release form, and HIPAA authorization form (or equivalent according to local regulations), reviewed and signed by the patient or legally authorized representatives.

Exclusion Criteria:

* Pediatric population and individuals under 50 years of age.
* Concomitant genetic musculoskeletal disorders.
* History of trauma.
* Spinal infections (spondylodiscitis, osteomyelitis, abscess, etc.).
* Presence of spinal tumors or other neoplasms.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 50-85 years) undergoing spinal surgery at the Fondazione Policlinico A. Gemelli IRCCS, a tertiary referral center specializing in neurosurgical care. Patients will be evaluated, assessed for surgical indication, and enrolled in the study at the Neurosurgery Department of the Institution.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Histological Modifications in the Ligamentum Flavum in Lumbar Spinal Stenosis and Other Degenerative Spinal Diseases | Intraoperative sample collection and subsequent laboratory analysis within 12 months post-surgery
  This outcome measures the relative abundance and structural organization of collagen and elastin fibers in ligamentum flavum tissue from patients with lumbar spinal stenosis and other degenerative spinal diseases, using histological staining.
  Unit of Measure: Histological score or percentage composition
Cellularity of Ligamentum Flavum Tissue | Intraoperative sample collection; analysis completed within 12 months post-surgery
  This outcome measures the number and density of fibroblasts and other resident cells in the ligamentum flavum.
  Unit of Measure: Cells per high power field (HPF)
Presence of Inflammatory Markers in Ligamentum Flavum | Intraoperative sample collection; analysis completed within 12 months post-surgery
  This outcome evaluates the expression of inflammatory markers (e.g., TNF-α, IL-6, CD68) in ligamentum flavum tissue using immunohistochemistry or immunofluorescence.
  Unit of Measure: Semi-quantitative histological score or intensity of staining

SECONDARY OUTCOMES:
Expression of Matrix Metalloproteinases (MMPs) in Ligamentum Flavum Tissue | Within 12 months post-surgery, based on sample processing and analysis.
  This outcome quantifies the expression of specific MMPs (e.g., MMP-2, MMP-9) involved in extracellular matrix remodeling in hypertrophied ligamentum flavum.
  Unit of Measure: Relative expression (e.g., fold-change via qPCR or densitometric units via Western blot)
Expression of Transforming Growth Factor-beta (TGF-β) in Ligamentum Flavum Tissue | Intraoperative tissue collection; laboratory analysis within 12 months post-surgery
  This outcome evaluates the expression of TGF-β, a key mediator in fibrosis and hypertrophy.
  Unit of Measure: Relative expression (e.g., immunohistochemistry score, qPCR fold-change)
Expression of Bone Morphogenetic Proteins (BMPs) in Ligamentum Flavum Tissue | Intraoperative tissue collection; laboratory analysis within 12 months post-surgery
  This outcome investigates the expression of BMPs (e.g., BMP-2, BMP-7) which are implicated in osteogenic changes and fibrosis.
  Unit of Measure: Relative expression (e.g., fold-change via qPCR or immunohistochemistry score)
Correlation Between Histological and Molecular Findings and Preoperative Clinical Presentation | Preoperative clinical data and intraoperative sample analysis; correlation analysis within 12 months
  This outcome assesses the relationship between tissue-based findings and clinical parameters such as pain, disability, and imaging severity.
  Unit of Measure: Correlation coefficient (e.g., Pearson's r or Spearman's ρ)
Correlation Between Histological and Molecular Findings and Postoperative Surgical Outcomes | Intraoperative sample collection and postoperative follow-up at 3, 6, and 12 months
  This outcome measures the association between tissue-level findings and surgical outcomes, including postoperative functional recovery (e.g., ODI, VAS, EQ5D).
  Unit of Measure: Correlation coefficient (e.g., Pearson's r or Spearman's ρ)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe La Rocca, Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCSS
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCSS, Rome, RM, Italy

REFERENCES:
- [Background] Zheng Z, Ao X, Li P, Lian Z, Jiang T, Zhang Z, Wang L. CRLF1 Is a Key Regulator in the Ligamentum Flavum Hypertrophy. Front Cell Dev Biol. 2020 Sep 18;8:858. doi: 10.3389/fcell.2020.00858. eCollection 2020. PMID 33072735
- [Background] Liu C, Li P, Ao X, Lian Z, Liu J, Li C, Huang M, Wang L, Zhang Z. Clusterin negatively modulates mechanical stress-mediated ligamentum flavum hypertrophy through TGF-beta1 signaling. Exp Mol Med. 2022 Sep;54(9):1549-1562. doi: 10.1038/s12276-022-00849-2. Epub 2022 Sep 21. PMID 36131026
- [Background] Wang AY, Saini H, Tingen JN, Sharma V, Flores A, Liu D, Olmos M, McPhail ED, Safain MG, Kryzanski J, Arkun K, Riesenburger RI. The Relationship Between Wild-Type Transthyretin Amyloid Load and Ligamentum Flavum Thickness in Lumbar Stenosis Patients. World Neurosurg. 2022 Aug;164:e113-e118. doi: 10.1016/j.wneu.2022.04.008. Epub 2022 Apr 6. PMID 35398327
- [Background] Zhao R, Dong J, Liu C, Li M, Tan R, Fei C, Chen Y, Yang X, Shi J, Xu J, Wang L, Li P, Zhang Z. Thrombospondin-1 promotes mechanical stress-mediated ligamentum flavum hypertrophy through the TGFbeta1/Smad3 signaling pathway. Matrix Biol. 2024 Mar;127:8-22. doi: 10.1016/j.matbio.2024.01.005. Epub 2024 Jan 26. PMID 38281553
- [Background] Troyer KL, Puttlitz CM. Nonlinear viscoelasticty plays an essential role in the functional behavior of spinal ligaments. J Biomech. 2012 Feb 23;45(4):684-91. doi: 10.1016/j.jbiomech.2011.12.009. Epub 2012 Jan 10. PMID 22236525
- [Background] Cheung PWH, Tam V, Leung VYL, Samartzis D, Cheung KM, Luk KD, Cheung JPY. The paradoxical relationship between ligamentum flavum hypertrophy and developmental lumbar spinal stenosis. Scoliosis Spinal Disord. 2016 Sep 5;11(1):26. doi: 10.1186/s13013-016-0088-5. eCollection 2016. PMID 27635416
- [Background] Lu QL, Wang XZ, Xie W, Chen XW, Zhu YL, Li XG. Macrophage migration inhibitory factor may contribute to hypertrophy of lumbar ligamentum flavum in type 2 diabetes mellitus. Chin Med J (Engl). 2020 Mar 5;133(5):623-625. doi: 10.1097/CM9.0000000000000680. No abstract available. PMID 31996548
- [Background] Tomkins-Lane CC, Battie MC, Hu R, Macedo L. Pathoanatomical characteristics of clinical lumbar spinal stenosis. J Back Musculoskelet Rehabil. 2014;27(2):223-9. doi: 10.3233/BMR-130440. PMID 24284271
- [Background] Katz JN, Zimmerman ZE, Mass H, Makhni MC. Diagnosis and Management of Lumbar Spinal Stenosis: A Review. JAMA. 2022 May 3;327(17):1688-1699. doi: 10.1001/jama.2022.5921. PMID 35503342
- [Background] Sobanski D, Staszkiewicz R, Stachura M, Gadzielinski M, Grabarek BO. Presentation, Diagnosis, and Management of Lower Back Pain Associated with Spinal Stenosis: A Narrative Review. Med Sci Monit. 2023 Feb 23;29:e939237. doi: 10.12659/MSM.939237. PMID 36814366